CLINICAL TRIAL: NCT07017348
Title: Knowledge and Exploratory Study to Better Understand the Gut-Skin Axis in Subjects With Moderate Atopic Dermatitis and Control Subjects
Brief Title: Assessment of Clinical, Biological and Biometrological Parameters in Adults Subjects With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GUTSKIN
Record Dates: First submitted 2025-05-14; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Atopic Dermatitis; Healthy
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control subject group (Other)
  Interventions: Other: Biometrological measurements; Other: Biological sampling; Other: Questionnaires
- Subject group with moderate atopic dermatitis (Other)
  Interventions: Other: Clinical assessments; Other: Biometrological measurements; Other: Biological sampling; Other: Questionnaires

INTERVENTIONS:
Other: Clinical assessments — dermatitis atopic scores will be evaluated on the entire body and on target areas by the investigator
  Arms: Subject group with moderate atopic dermatitis
Other: Biometrological measurements — Measurements will be performed on the target areas
Other: Biological sampling — Skin and faecal samples will be performed
Other: Questionnaires — dietary habits, health and lifestyle, and digestive health

SUMMARY:
In most recent years, the gut microbiome has been highlighted as a key player in the control of organs distant from the gut. Indeed, studies have raised evidence that gut microbiota exerts a control on various diseases including joint, cardiovascular, metabolic, or skin diseases, and even mental health.

Many of these effects are attributed to the role of microbiota in controlling intestinal mucosa immunity. For skin diseases, and in particular for Atopic Dermatitis (AD), it has been suggested that the imbalance of the gut microbiome affects systemic inflammation and immune response, which leads to an exacerbation of AD. Complementary to a gut-driven activation of systemic immunity, a role for the nervous system, or even for hormonal pathways can also be envisioned as contributors to the effects of gut microbiome on AD.

Understanding how the gut microbiome controls skin biology, whether it involves or not the immune system, still requires extensive translational research. A better knowledge of the actors and markers of the Gut-Skin axis is therefore necessary to understand the exact mechanisms by which the gut microbiome influences or aggravates AD symptoms.

The study will be conducted in adult subjects, divided into 2 groups:

* Group AD: subjects with moderate atopic dermatitis
* Group CTRL: subjects with no inflammatory dermatological pathology

Number of visits:

2 visits maximum are planned for both groups:

* Visit 1: Inclusion ± end-of-study visit (Day 1)
* Collection phase at home*: 1 to 5 days (Day 1 to Day 6)
* Visit 2**: End-of-study visit (Day 2 to Day 6) (maximum 24h after faecal sampling at home)

  * If faecal sampling was not possible during the inclusion visit, the kit will be kept by the subject to collect the sample at home.

    * Only if the faecal sampling is carried out at home.

The maximal duration of participation for a subject is 6 days from the inclusion visit to the end of the study.

ELIGIBILITY:
Inclusion criteria

Criteria related to the population:

* Female
* Subject aged of 18 years old and over
* Subject non-menopausal
* For woman of childbearing potential:

  * use of an effective method of contraception, as assessed by the investigator, introduced and unchanged for at least 1 month before inclusion in the study
  * accept to go on using it during the whole duration of the study

Criteria related to the diseases and/or skin conditions:

Specific for the AD group:

* Subject with atopic dermatitis according to "The U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis"
* Subject with moderate atopic dermatitis with a SCORAD between 25 and 40 included
* Subject with target areas on the upper or lower limbs allowing sampling and measurements, defined as:

  * Area of usual atopic dermatitis flare-up with at least one inflammatory flare-up of AD in the year preceding the inclusion visit
  * Area not in actual flare-up but with the following L-SCORAD signs (18-point scale):

    * Erythema score ≥ 1 on a scale ranged from 0 to 3
    * Xerosis score ≥ 1 on a scale ranged from 0 to 3

Specific for the CTRL group:

Subject without inflammatory dermatological conditions (skin and scalp)

Non-inclusion criteria

Criteria related to the population:

* For woman of childbearing potential: pregnant or breastfeeding or planning to be pregnant during the study
* Subject having received on target areas artificial UV exposure, excessive or prolonged exposure to natural sunlight within 2 weeks before the inclusion visit
* Subject hirsute on the target areas
* Subject who has shaved or waxed the target areas within the last 2 days before the inclusion visit

Criteria related to the diseases and/or skin conditions:

* Subject having a dermatological condition (excepted AD for atopic dermatitis group), an acute, chronic or progressive disease or history of disease liable to interfere with the study data or considered by the investigator hazardous for the subject or incompatible with the study requirements
* Subject having any other dermatologic condition than atopic dermatitis (for AD group), or characteristics (like tattoo) on the target areas liable to interfere with the study assessments according to the judgement of the investigator
* Subject with intestinal diseases or food allergies liable to interfere with the study, in the opinion of the investigator

Specific for the atopic dermatitis group:

* Subject with a flare-up of AD (requiring a topical or systemic medical treatment in the opinion of the investigator)
* Subject with superinfected AD

Criteria related to treatments and/or products:

* Systemic immunosuppressive treatment (except corticosteroids) taken within 3 months before the inclusion visit or planned during the study
* Systemic antibiotics treatment taken within 4 weeks before the inclusion visit or planned during the study
* Dietary supplements or probiotics taken within 4 weeks before the inclusion visit or planned during the study
* Systemic corticosteroids treatment taken within 4 weeks before the inclusion visit or planned during the study
* Laxative taken within 4 weeks before the inclusion visit or planned during the study
* Phototherapy within 4 weeks before the inclusion visit or planned during the study
* Colonoscopy within 4 weeks before the inclusion visit or planned during the study
* Systemic treatment with NSAID taken in the 7 days prior to the inclusion visit or ongoing at the inclusion visit (from 3 days of intake)
* Topical corticosteroids treatment applied on target areas within 7 days before the inclusion visit or planned during the study
* Topical immunomodulating treatment applied on target areas within 7 days before the inclusion visit or planned during the study
* Topical treatment with NSAID applied on target areas within 7 days before the inclusion visit or planned during the study
* Topical emollient applied on target areas within the last 48h before the inclusion visit
* Any treatment, topical product (excepted emollient) and/or water applied on target areas between the last shower (maximum the evening before inclusion visit) and the inclusion visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Atopic dermatitis severity on the entire body | baseline (Visit 1- Day 1)
  by SCORAD on a scale 0 to 103 in atopic dermatitis group only
Atopic dermatitis severity on target areas | baseline (Visit 1- Day 1)
  by L-SCORAD on a scale 0 to 18 in atopic dermatitis group only
Cutaneous pH measurement | baseline (Visit 1- Day 1)
  by pH - pHmeter
Cutaneous hydration | baseline (Visit 1- Day 1)
  by Hydration Index (IH) - Corneometer®
Cutaneous barrier integrity | baseline (Visit 1- Day 1)
  by Trans-Epidermal Water Loss (TEWL) - Vapometer®
Microbiota analysis by sampling method with swab by gene sequencing data | baseline (Visit 1- Day 1)
Microbiota analysis by sampling method with feces by gene sequencing data | baseline (Visit 1- Day 1, or Visit 2 - Day 2 to 6)
Metabolites analysis by sampling method with swab by metabolomic technics with mass spectrometry | baseline (Visit 1- Day 1)
Metabolites analysis by sampling method with feces by metabolomic technics with mass spectrometry | baseline (Visit 1- Day 1, or Visit 2 - Day 2 to 6)
Lipids analysis by sampling method with swab by absolute quantification with mass spectrometry | baseline (Visit 1- Day 1)
Proteins analysis by sampling method with feces by metaproteomics workflow with mass spectrometry | baseline (Visit 1- Day 1, or Visit 2 - Day 2 to 6)
Proteins analysis by sampling method with swab by metaproteomics workflow with mass spectrometry | baseline (Visit 1- Day 1)
Digestive health by a questionnaire in both groups on digestive discomfort and abdominal pain | baseline (Visit 1- Day 1)
Dietary habits, health and life by a questionnaire in both groups on diet, consumption of foods, health and lifestyle | baseline (Visit 1- Day 1)
Illustrative photographs of target areas in atopic dermatitis group only | baseline (Visit 1- Day 1)
  The standardized photographs of target areas in the atopic dermatitis group are intended solely for illustrative purposes. They do not serve as a quantitative measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Research Center, Toulouse, France